CLINICAL TRIAL: NCT07094958
Title: Efficacy of Intradermal Stromal Vascular Fraction Injection in the Treatment of Atrophic Acne Scar
Brief Title: Efficacy of Stromal Vascular Fraction on Acne Scar Correction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Acne scar_SVF study
Record Dates: First submitted 2025-07-29; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Acne Scars; Acne Scars - Atrophic
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVF-treated side (Experimental): Intradermal injection of autologous stromal vascular fraction (SVF) on one side of the face.
  Interventions: Biological: stromal vascular fraction (SVF)
- Saline-treated side (Placebo Comparator): Intradermal injection of normal saline (NS) on the contralateral side of the face.
  Interventions: Other: Normal Saline (NS)

INTERVENTIONS:
Biological: stromal vascular fraction (SVF) — Autologous stromal vascular fraction (SVF) isolated from adipose tissue was injected intradermally into one side of the face to evaluate its efficacy in treating atrophic acne scars. SVF was freshly prepared on the same day of injection using enzymatic digestion and centrifugation.
  Arms: SVF-treated side
Other: Normal Saline (NS) — Normal saline (NS) was injected intradermally into the contralateral side of the face and served as a placebo comparator to SVF in this split-face study on atrophic acne scars.
  Arms: Saline-treated side

SUMMARY:
This study aims to evaluate the efficacy and safety of intradermal injection of autologous stromal vascular fraction (SVF) in the treatment of atrophic acne scars. SVF is a heterogeneous cell population derived from adipose tissue, containing various regenerative and immunomodulatory cells, including mesenchymal stem cells, endothelial progenitor cells, and pericytes.

In this prospective, randomized, split-face clinical trial, participants with atrophic acne scars will receive SVF injections on one side of the face and normal saline (NS) injections on the contralateral side as a control. Clinical efficacy will be assessed through blinded scar counts, digital imaging, and histological evaluations including epidermal and dermal regenerative markers. The study is designed to investigate whether SVF provides superior clinical improvement compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 45 years
* Presence of bilateral atrophic acne scars (boxcar, rolling, or icepick types) on the face
* Willingness to undergo fat harvesting procedure
* Ability to comply with study visits and follow-up
* Written informed consent obtained

Exclusion Criteria:

* Active acne lesions on the treatment area
* History of keloid or hypertrophic scarring
* Prior treatment for acne scars (e.g., laser, filler, microneedling) within the past 6 months
* History of systemic immunosuppressive therapy within the past 3 months
* Pregnant or breastfeeding women
* Any systemic disease that may interfere with wound healing or safety assessment (e.g., uncontrolled diabetes, collagen vascular disease)

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in total number of atrophic acne scars from baseline to Week 5 | Baseline and 5 weeks after treatment
Change in total number of atrophic acne scars from baseline to Week 10 | Baseline and 10 weeks after treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mbiine R, Wayengera M, Kiwanuka N, Munabi I, Muwonge H, Nakanwagi C, Joloba M, Galukande M. Autologous adipose-derived stromal vascular fraction (SVF) in scar treatment among patients with keloids and hypertrophic scars: a systematic review and meta-analysis of current practices and outcomes. Am J Stem Cells. 2023 Dec 15;12(5):98-111. eCollection 2023. PMID 38213639
- [Background] Bora P, Majumdar AS. Adipose tissue-derived stromal vascular fraction in regenerative medicine: a brief review on biology and translation. Stem Cell Res Ther. 2017 Jun 15;8(1):145. doi: 10.1186/s13287-017-0598-y. PMID 28619097
- [Background] Connolly D, Vu HL, Mariwalla K, Saedi N. Acne Scarring-Pathogenesis, Evaluation, and Treatment Options. J Clin Aesthet Dermatol. 2017 Sep;10(9):12-23. Epub 2017 Sep 1. PMID 29344322
- [Background] Dreno B, Layton A, Bettoli V et al. Evaluation of the prevalence, risk factors, clinical characteristics, and burden of acne scars among active acne patients in brazil, france, and the USA. J Am Acad Dermatol 2017; 76:ab132.
- [Background] Kwon HH, Yoon HS, Suh DH, Yoon JY, Park SK, Lee ES, Lee JH, Kim NI, Kye YC, Ro YS, Lee SJ, Kim MN, Sung KJ, Lee ES, Kim KJ; Korean Society for Acne Research. A nationwide study of acne treatment patterns in Korea: analysis of patient preconceived notions and dermatologist suggestion for treatment. Acta Derm Venereol. 2012 May;92(3):236-40. doi: 10.2340/00015555-1331. PMID 22367348
- [Background] Eichenfield DZ, Sprague J, Eichenfield LF. Management of Acne Vulgaris: A Review. JAMA. 2021 Nov 23;326(20):2055-2067. doi: 10.1001/jama.2021.17633. PMID 34812859
- [Derived] Suh JH, Kim JY, Yoon JY, Lee JH, Kim DH, Jin U, Suh DH. Comparison of Efficacy of Intradermal Stromal Vascular Fraction Injection Versus Saline Injection in the Treatment of Atrophic Acne Scar: A 10-Week, Prospective, Randomized, Split-Face, Single-Blind Controlled Trial. Dermatol Ther (Heidelb). 2025 Dec 18. doi: 10.1007/s13555-025-01617-6. Online ahead of print. PMID 41413319